CLINICAL TRIAL: NCT06760312
Title: Effect of Different Apical Actions on Local Inflammatory Mediators and Pain During Root Canal Preparation: A Randomized Clinical Study
Brief Title: Effect of Different Apical Actions on Local Inflammatory Mediators and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Emrah Karataşlıoğlu, Associate Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-KAE-0080
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Dental Pain; Pulp Disease, Dental; Pulpitis - Irreversible
Keywords: apical kinematics; apical action; apical reverse; apical slow-down; continuous rotation; Substance P; postoperative pain; Inflammation
MeSH Terms: conditions — Dental Pulp Diseases; Pain, Postoperative; Inflammation

STUDY DESIGN:
Intervention Model Description: n=66 participants will be randomized into 3 different intervention groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuous Rotation (Experimental): The apical root canal shaping mode of the apex locator integrated endodontic motor is "Continuous Rotation" which is the standard and mostly used option in endodontics. Works as a Control group also
  Interventions: Procedure: Root canal shaping with Continuous Rotation
- Apical Reverse (Experimental): The apical root canal shaping mode of the apex locator integrated endodontic motor is "Reverse". The motor makes a reverse movement to prevent the file over the working length
  Interventions: Procedure: Root canal shaping with Apical Reverse
- Apical Slow-down (Experimental): The apical root canal shaping mode of the apex locator integrated endodontic motor is "Apical Slow-down". The motor slows down the rotation to preserve the working length and apical constriction.
  Interventions: Procedure: Root canal shaping is conducted with Apical slow-down kinematic.

INTERVENTIONS:
Procedure: Root canal shaping with Continuous Rotation — The root canal shaping is conducted with a continuous rotation kinematic.
  Arms: Continuous Rotation
Procedure: Root canal shaping with Apical Reverse — The root canal shaping is conducted with a apical reverse kinematic.
  Arms: Apical Reverse
Procedure: Root canal shaping is conducted with Apical slow-down kinematic. — The root canal shaping is conducted with a apical slow-down kinematic.
  Arms: Apical Slow-down

SUMMARY:
The goal of this clinical trial is to determine patients' the inflammation and pain response to different apical actions used in rotary instrumentation during root canal shaping process. The main questions it aims to answer are:

1. How the different apical actions of endodontic motors influence the pain and inflammatory mediator release from the periapical region of related tooth?
2. Does the perceived pain differ among the used apical action methods after the root canal preparation?
3. Are the perceived pain and local pain mediator levels coherent?

Participants will:

Attend to the root canal treatment in the endodontics clinic. The treatment will be two visits.

Answer the Visual Analog Scale questionnaire on day 0 (first appt.) and Day 3 (second appt.) Keep a diary of their symptoms and the number of times they use an anti-inflammatory drug.

DETAILED DESCRIPTION:
Study Protocol

This study will include patients aged 18-49 years who present to the İzmir Katip Çelebi University, Department of Endodontics, requiring root canal treatment for vital, lesion-free mandibular first and second molars. Patients with systemic diseases will be excluded. The study will involve 66 patients. The sample size was calculated according to the effect size of 0,25 recommended by Cohen (1988).

Pre-Treatment Assessment:

* Patients will be asked about spontaneous pain and percussion pain related to the affected tooth prior to the session.
* These pain levels will be recorded using the Visual Analog Scale (VAS).

Group Allocation:

* After rubber dam isolation and access cavity preparation, patients will be randomly assigned to one of four groups using a four-sided die.
* Each group will consist of 22 patients and will undergo root canal shaping using an endomotor with one of the following techniques:

  1. Continuous Rotation
  2. Apical Reverse
  3. Apical Slow-Down

Questionnaire:

Patients will be given a pen and will be asked to mark the current and percussion-provoked pain of the related tooth by a numbered linear Visual Analog Scale (VAS) before treatment on Day 0 and Day 3.

Root Canal Shaping:

1. Working Length Determination: Establish the working length and create a glide path using a #10 K-file.
2. Instrumentation Sequence: Enlarge the canals sequentially using rotary files of sizes 15.04, 20.04, 25.06, 30.06, and 35.06.
3. Irrigation: Use 2 ml of 2.5% sodium hypochlorite (NaOCl) for irrigation after each file change.

Sample Collection (First Session):

* After completing the first session:
* Rinse the canals with distilled water.
* Remove remaining liquid with #45 paper points.
* Insert sterile #20.02 paper points into the canals and leave them for 30 seconds to collect periapical exudates.
* Collect three samples per canal. Cut the apical 5 mm of the paper points and place them in 1.5 ml Eppendorf tubes for storage at -80°C.
* The canals will then be rinsed again with 2.5% NaOCl. Patients will be dismissed without using intra-canal medication and instructed to return for the filling session after three days. Patients will be advised to take 800 mg ibuprofen if they experience pain. The medication use will be documented.

Second Session:

* The questionnaire will be held again with the VAS scores and percussion sensivity.

  * After local anesthesia the intermediate restorative material is removed and root canal irrigation with distilled water.
  * Working length is confirmed again with a file. Collect three additional samples per canal using #20.02 paper points as in the first session.
  * Proceed to finalize the root canal treatment.

Final Root Canal Treatment:

1. Perform the final irrigation using 2.5% sodium hypochlorite and 17% EDTA.
2. Fit gutta-percha cones. 35.06 cone or fitting .02 tapered cones will be selected as the master cone according to the anatomy and fit.
3. Fill the canals using a resin-based root canal sealer with lateral condensation utilizing #25 spreader and accessory #20.02 gutta-percha cones.
4. After cutting the excess gutta-percha, clean the cavity and complete the treatment with composite resin restoration.

Sample Handling:

* All collected samples will be stored in a -80°C freezer for biochemical analysis. The analysis will be based on ELISA tests which will investigate the Substance P, IL-1ß, TNF alpha and IL-6 on Day 0 and Day 3.

Post-Treatment:

* The occlusion will be checked using articulation paper, and adjustments will be made if primary contact is present to ensure no traumatic occlusion.

This standardized protocol ensures consistent data collection and optimal treatment outcomes for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate pulpitis and pulpal expose patients in need of root canal -treatment to their mandibular premolars.
* Healthy periodontal tissue with Periapical Index under 2.
* Helathy adjacent teeth.

Exclusion Criteria:

* Systemic diseases
* Percussion pain
* Patients who did not consent to a vital pulp therapy
* Radiologically seen open apex, root resorption, calcification
* Periodontal pocket beyond 4mm in length
* Consumption of Antibiotics or Corticosteroids 1 month before the treatment
* Consumption of antiinflammatory drugs 2 days before the treatment

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Substance P | From Day 0 to Day 3. The last measurement will be taken just before the end of the interventional treatment.
  The local Substance P amount will be assesed with ELISA kits

SECONDARY OUTCOMES:
Visual Analog Scale | From Day 0 to Day 3. The last measurement will be taken just before the end of the interventional treatment.
  Visual Analog Scale (VAS) questionnaire of perceived pain. A visual linear scale starting from 0 to 10. 0 represents no pain and 10 is the highest pain patient ever endured. Patient is asked to mark the pain in the scale.
Inflammatory Mediator: IL-1ß | From Day 0 to Day 3. The last measurement will be taken just before the end of the interventional treatment.
  Local IL-1ß will be assessed with local collection from apical site.
Inflammatory Mediator: IL-6 | From Day 0 to Day 3. The last measurement will be taken just before the end of the interventional treatment.
  Local IL-6 will be assessed with local collection from apical site.
Inflammatory Mediator: TNF alpha | From Day 0 to Day 3. The last measurement will be taken just before the end of the interventional treatment.
  Local TNF-alpha will be assessed with local collection from apical site.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Karataşlıoğlu, PhD, Study Chair — İzmir Katip Çelebi Üniversitesi; Mustafa Mert Tulgar, Dmd, Principal Investigator — İzmir Katip Çelebi Üniversitesi; Yağmur Kılıç, Dmd, Principal Investigator — İzmir Katip Çelebi Üniversitesi
Locations (1):
- İzmir Katip Çelebi Üniversitesi, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The patients' written consent also required that the data, which involves biological markers, be used only within the experiment and not shared with a third party.

REFERENCES:
- [Background] Cohen, J (1988) Statistical power analysis for the behavioral sciences (2nd ed.). Hillsdale, NJ: Erlbaum